CLINICAL TRIAL: NCT07383207
Title: The Effect of Problem-Based Microlearning on Nursing Students' Knowledge Level, Self-Directed Learning, and Reflective Thinking Skills Regarding Movement Requirements: A Randomized Controlled Trial
Brief Title: Microlearning and the Requirement for Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Aysun Acun 13
Record Dates: First submitted 2025-11-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-11

CONDITIONS: Nursing Students
Keywords: Microlearning; movement; problem-based learning

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nursing students (Experimental): Nursing students' knowledge level
  Interventions: Other: knowledge level

INTERVENTIONS:
Other: knowledge level — The Effect of Problem-Based Microlearning on Nursing Students' Knowledge Level

SUMMARY:
This research aims to explain the effect of problem-based micro learning on nursing students' knowledge level, self-directed learning, and reflective thinking skills regarding the need for movement.

DETAILED DESCRIPTION:
This study aims to use problem-based microlearning strategies in an integrated manner so that students can comprehend information in depth rather than just superficially and use this information effectively in a clinical setting. The application of problem-based micro learning to first-year nursing students regarding the need for movement constitutes the original aspect of the study. The research is expected to contribute to the literature in terms of the development of knowledge-based skills such as positioning patients, safe transfer, and joint mobilization movements.

ELIGIBILITY:
Inclusion Criteria:

* Not having previously received training on movement requirements knowledge and skills
* Course attendance, participation in the final test and follow-up test

Exclusion Criteria:

* Previously having received training on movement requirements knowledge and skills
* Absence from class, not participating in the final test and follow-up test
* Students who have difficulty speaking and understanding Turkish

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Nursing students
Enrollment: 105 (Actual)
Dates: Start 2025-11-20 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Information test on movement requirements (20 questions) | 7 weeks
  Nursing students' knowledge level

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Bilecik, Turkey (Türkiye)